CLINICAL TRIAL: NCT05613010
Title: Leveraging Technology to Improve Medication Adherence in Adolescent and Young Adult Kidney or Liver Transplant Recipients: A Micro-Randomized Trial
Brief Title: Leveraging Technology to Improve Medication Adherence in Youth With Kidney or Liver Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00321009; K23DK128573 (NIH)
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Transplant;Failure,Kidney; Transplant; Failure, Liver; Adherence, Medication; Adherence, Patient; Adherence, Treatment
Keywords: kidney transplant; liver transplant; medication adherence; medication nonadherence; compliance; mobile health; mobile phone; technology
MeSH Terms: conditions — Medication Adherence; Patient Compliance; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This study uses a within-subjects micro-randomized trial design. This study involves randomizing participants within person hundreds of times over to receive intervention or not at each expected dose. Each dose is a decision-point to deliver intervention or not, allowing for within-person comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile health (mHealth) text messaging intervention (Experimental): During baseline (4 weeks), adherence will be monitored daily via electronic pill boxes and no text messages will be sent. After baseline, participants will begin the 12-week micro-randomized trial of the intervention (a within-person study design). During this 12-week micro-randomized trial, daily adherence will be electronically monitored with the electronic pill boxes and participants will be randomized to receive (1) adherence support text messages or (2) no text message after each missed dose, and (1) praise text message or (2) no text message after each on time dose. For 12 months post-intervention, participants will keep using the electronic pill boxes (no text messages will be sent).
  Interventions: Behavioral: mHealth Messaging Intervention Group

INTERVENTIONS:
Behavioral: mHealth Messaging Intervention Group — Participants will receive an electronic pill box; the research team will instruct participants on how to use this device. Participants will be asked to use the electronic pill box for their prescribed medicines for the duration of the study (up to 16 months). During the 12-week micro-randomized trial, participants will be randomized within person to receive (1) adherence support text messages or (2) no text message after each missed dose, and (1) praise text message or (2) no text message after each on time dose. Dose timing will be determined based on participant report of when they typically take their tacrolimus or sirolimus medicine.

SUMMARY:
Can the investigators create an effective way to improve adherence to immunosuppressant medication and reduce rejection, graft loss, and death in adolescents and young adults who have undergone kidney or liver transplantation? The investigators' mobile technology intervention uses real-time electronic pillbox-assessed dose timing and text message prompts to address antirejection medication nonadherence when nonadherence is detected.

DETAILED DESCRIPTION:
Over 1/3 of adolescents and young adults who have undergone kidney or liver transplantation are nonadherent to antirejection medicines, accounting for shockingly high rates of infections, rejection, graft loss, and even death. Recently, the American Society of Transplantation highlighted real-time adherence intervention as top priorities to address antirejection medication nonadherence, but these evidence-based intervention tools do not exist. The investigators aim to answer the American Society of Transplantation's call and fill these critical gaps in nonadherence management for adolescents and young adults with kidney or liver transplant. Specifically, electronic pillboxes yield valuable real-time daily dosing data to guide interventions for adolescents and young adult kidney or liver transplant recipients, but existing interventions have not optimally leveraged these devices' capabilities. Just-in-time adaptive interventions delivered via mobile device (i.e., Smartphone or tablet) are cutting-edge approaches that fully incorporate adolescents and young adults' daily dose behavior to automatically deliver tailored intervention content exactly when adolescents and young adults need it most. The investigators piloted a promising static medication adherence support text message intervention based on the COM-B model, a well-established behavioral health intervention model, which will be modified into a just-in-time adaptive intervention for adolescents and young adult kidney or liver transplant recipients. Given that 95% of adolescents and young adults in the USA own smartphones, the investigators hypothesize that the investigators' intervention will improve on-time dosing and reduce rejection, graft loss, and death. The investigators believe that providing adherence support text messages or praise text messages will result in a higher proportion of adolescents and young adults taking the next dose and maintaining improvements in adherence post-intervention. In summary, the investigators' just-in-time adaptive intervention leverages real-time electronic pillbox-assessed dosing behavior and Smartphone text messaging capabilities to address tacrolimus or sirolimus nonadherence when nonadherence is detected.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults (13-25 years old) who underwent kidney or liver transplantation at least 6 months prior to enrollment
* Currently prescribed tacrolimus or sirolimus.

Exclusion Criteria:

* Currently receiving dialysis
* Hospitalized for duration of study
* Significant developmental or cognitive delay
* No access to a mobile device that supports text messaging
* Decline to use electronic pill box to monitor daily medication adherence
* Non-English speaking
* If a participant meets inclusion criteria, enrolls in the study, and experiences graft failure potentially leading to dialysis in the case of kidney transplant recipients, the participant will be given the option to continue in the study if they remain on tacrolimus or sirolimus.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Electronically-measured medication adherence (dose taken or not) | 16 months
  Participants will use an electronic pillbox to assess daily immunosuppressant adherence (tacrolimus or sirolimus), defined as a binary variable: dose taken or not.

SECONDARY OUTCOMES:
Standard deviation of antirejection medication dose timing | 16 months
  This metric will be calculated as each participants' standard deviation (SD) in tacrolimus or sirolimus daily dose timing during the study based on how many minutes early/late tacrolimus or sirolimus was timestamped as taken (administered) from when it is prescribed (e.g., how many minutes before/after AYA's expected dose time) using time stamp data from the electronic pill boxes.

CONTACTS AND LOCATIONS:
Overall Officials: Cyd Eaton, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be shared in a de-identified form (i.e., clean, de-identified electronic database) upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon request
Access Criteria: Data from this study will be shared in a de-identified form (i.e., clean, de-identified electronic database).